CLINICAL TRIAL: NCT05972044
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Trial of Solriamfetol in Adults With ADHD.
Brief Title: A Study to Assess the Efficacy and Safety of Solriamfetol in Subjects With ADHD (FOCUS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOL-ADHD-301
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: ADHD
Keywords: Attention deficit hyperactivity disorder; ADHD; Solriamfetol; Sunosi; Axsome; Non-stimulant therapy; Dopamine norepinephrine reuptake inhibitor
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — solriamfetol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Solriamfetol 150 mg (Experimental): Up to 6 weeks
  Interventions: Drug: Solriamfetol 150 mg
- Solriamfetol 300 mg (Experimental): Up to 6 weeks
  Interventions: Drug: Solriamfetol 300 mg
- Placebo (Placebo Comparator): Up to 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solriamfetol 150 mg — Solriamfetol tablets, taken once daily
  Arms: Solriamfetol 150 mg
Drug: Solriamfetol 300 mg — Solriamfetol tablets, taken once daily
  Arms: Solriamfetol 300 mg
Drug: Placebo — Placebo tablets, taken once daily
  Arms: Placebo

SUMMARY:
FOCUS (Forward Treatment of Attention Deficit and Hyperactivity Using Solriamfetol) is a Phase 3, multi-center, randomized, double-blind, placebo-controlled, parallel- group trial to assess the efficacy and safety of solriamfetol in adults with ADHD.

DETAILED DESCRIPTION:
Eligible subjects must have a primary diagnosis of ADHD based on the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM-5) criteria. Subjects will be randomized in a 1:1:1 ratio to be treated with solriamfetol 150 mg, solriamfetol 300 mg, or placebo, once daily for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of ADHD according to DSM-5 criteria.
* Provides written informed consent to participate in the study before the conduct of any study procedures.
* Male or female, aged 18 to 55 inclusive.

Exclusion Criteria:

* Prior exposure to solriamfetol/Sunosi, through either a clinical study or prescription.
* Unable to comply with study procedures.
* Medically inappropriate for study participation in the opinion of the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 516 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 6 in the AISRS total score | 6 weeks
  Adult ADHD Investigator Symptom Report Scale (AISRS)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (40):
  - Clinical Research Site, Encino, California
  - Clinical Research Site, Garden Grove, California
  - Clinical Research Site, Newport Beach, California
  - Clinical Research Site, Riverside, California
  - Clinical Research Site, Santa Ana, California
  - Clinical Research Site, Sherman Oaks, California
  - Clinical Research Site, Torrance, California
  - Clinical Research Site, Walnut Creek, California
  - Clinical Research Site, Colorado Springs, Colorado
  - Clinical Research Site, Clermont, Florida
  - Clinical Research Site, Doral, Florida
  - Clinical Research Site, Gainesville, Florida
  - Clinical Research Site, Jacksonville, Florida
  - Clinical Research Site, Lauderhill, Florida
  - Clinical Research Site, Miami Lakes, Florida
  - Clinical Research Site, Orlando, Florida
  - Clinical Research Site, Marietta, Georgia
  - Clinical Research Site, Overland Park, Kansas
  - Clinical Research Site, Boston, Massachusetts
  - Clinical Research Site, Saint Charles, Missouri
  - Clinical Research Site, Lincoln, Nebraska
  - Clinical Research Site, Las Vegas, Nevada
  - Clinical Research Site, Berlin, New Jersey
  - Clinical Research Site, Cherry Hill, New Jersey
  - Clinical Research Site, Princeton, New Jersey
  - Clinical Research Site, Mount Kisco, New York
  - Clinical Research Site, New York, New York
  - Clinical Research Site, Raleigh, North Carolina
  - Clinical Research Site, Cincinnati, Ohio
  - Clinical Research Site, Kettering, Ohio
  - Clinical Research Site, Oklahoma City, Oklahoma
  - Clinical Research Site, Media, Pennsylvania
  - Clinical Research Site, North Charleston, South Carolina
  - Clinical Research Site, Memphis, Tennessee
  - Clinical Research Site, Austin, Texas
  - Clinical Research Site, Bellaire, Texas
  - Clinical Research Site, Dallas, Texas
  - Clinical Research Site, San Antonio, Texas
  - Clinical Research Site, Draper, Utah
  - Clinical Research Site, Everett, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Axsome Therapeutics Website — http://www.axsome.com